CLINICAL TRIAL: NCT06019871
Title: Danish Cohort for Patients Over 75 Years of Age With Chronic Kidney Disease Stage Five Who Are on Dialysis Treatment or on a Conservative Kidney Management Pathway
Brief Title: The Danish Symptomburden Study Among Patients With Advanced Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 15032023
Record Dates: First submitted 2023-03-06; First posted 2023-08-31 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decided for conservative kidney management: Patient with advanced kidney disease and decided for conservative kidney management
- Decided for dialysis: Patient with advanced kidney disease and decided for dialysis
  Interventions: Procedure: Dialysis

INTERVENTIONS:
Procedure: Dialysis — Patients who have decided for dialysis either center haemo-dialysis or peritoneal dialysis
  Groups: Decided for dialysis

SUMMARY:
Patients with chronic kidney disease stage five have a high symptom burden regardless of whether they are treated with dialysis or without dialysis, a conservative kidney management pathway (CKM). Previously, there has not been a validated tool in Danish to collect information about symptoms. The Integrated Palliative Outcome Scale Renal (IPOS-Renal) has now been validated and translated into Danish. IPOS-Renal aims to identify symptoms among patients with chronic kidney disease stage five.

The purpose of the study is to investigate whether there is a correlation between treatment - dialysis (haemodialysis or peritoneal dialysis) or CKM for patients >75 years of age with chronic kidney disease stage V and their symptom burden measured with IPOS-Renal. In addition, it is investigated whether there is a correlation between treatment - dialysis or CKM for patients >75 years of age with chronic kidney disease stage V and their mortality.

The study will be conducted as an observational prospective cohort study over a two-year period, and based on a power calculation, it is expected to include 341 patients with data originating from 11 hospitals in Denmark. Comparison of change in symptom burden over time measured by IPOS-Renal for the two forms of treatment will be examined as continuous data, and then the t-test or Mann-Whitney test will be used. A cox proportional hazard regression analysis will be used to examine mortality for patients in dialysis treatment and patients on CKM pathway.

DETAILED DESCRIPTION:
Background In chronic kidney disease stage five, patients must decide whether they want to start treatment with dialysis or a conservative kidney management pathway (CKM). It is a major decision for patients and their relatives, which concerns survival, quality of life, symptom burden and time spent in hospital. Patients with chronic kidney disease stage five have a high symptom burden, regardless of whether they are treated with dialysis or on CKM pathway. Systematic observation and recording of the symptoms should take place and alleviated to the extent possible. The patients experience a number of different symptoms including fatigue, nausea, dyspnoea, reduced level of physical function, pain and restlessness in the legs. A systematic review based on 25 primary studies found that there is an increased mortality in patients on an CKM pathway compared to patients on dialysis. But at the same time, benefits are seen in relation to increased quality of life, reduced symptom burden and fewer hospitalizations if the patient is on CKM pathway. Another study reports that patients in dialysis treatment have a higher symptom burden, lower well-being and poorer quality of life than patients who have opted out of dialysis.

In Denmark, symptoms experienced by patients with chronic kidney disease stage five are not systematically recorded, as there has not previously been a tool to collect Patient Reported Outcomes . The Integrated Palliative Outcome Scale Renal (IPOS-Renal) for patients with chronic kidney disease stage five is a validated screening tool to systematically investigate which symptoms patients with chronic kidney disease stage five report. Routinely collecting data about the patient's symptoms is the first step to improve care and treatment for patients with stage five chronic kidney disease. The validation and translation of the Danish IPOS-Renal was carried out in 2019-2020 by principal investigator. The implementation of IPOS-Renal can help to provide an increased focus on symptom management and quality of life among patients with chronic kidney disease stage five. IPOS-Renal gives patients the opportunity to be further involved in their disease and health, as the patients themselves have the opportunity to complete the questionnaire. IPOS-Renal takes less than 10 minutes to complete. IPOS-Renal contains a total of 11 questions concerning the most common physical symptoms for patients with chronic kidney failure. In addition, IPOS-Renal also contains questions about the patient's mental and existential needs, social needs and practical needs.

Purpose The purpose of the current study is to investigate whether there is a correlation between patients >75 years of age with chronic kidney disease stage five in treatment with - dialysis or on a CKM pathway and their symptom burden measured with the IPOS-Renal score. In addition, it is investigated whether there is a correlation between patients >75 years of age with chronic kidney disease stage five in treatment with - dialysis or on a CKM pathway and their mortality.

Hypotheses I. Patients on a CKM pathway have greater improvement in their symptom burden measured with IPOS-Renal than patients in dialysis treatment. II. Patients in dialysis treatment have a lower mortality rate than patients on a CKM pathway.

Materials and methods The project will be carried out as an observational prospective cohort study of patients with chronic kidney disease stage five in dialysis treatment or on a CKM pathway. Data originate from patients from 11 hospitals in Denmark: Aalborg University Hospital, Regionshospitalet Gødstrup, Sydvestjysk Sygehus, Kolding Hospital, Gegehus Sønderjylland Sønderborg, Rigshospitalet, Sjællands University Hospital Roskilde, Nykøbing Falster Hospital, Herlev Hospital, North Zealand Hospital and Aarhus University Hospital. In the current study, baseline information is defined at the patient's first response to the questionnaire. After that, the questionnaire is answered every 6 months for two years or until death.

Study population The patients will be included right after they have made their decision about treatment - dialysis (haemodialysis or peritoneal dialysis) or CKM pathway. In addition, patients must meet inclusion criteria. The patients will be observed for at least two years or until death. The study started on 15.03.2023, and it is expected to be completed on 14.03.2025.

Data collection and procedure All patients who meet the inclusion criteria and have chosen treatment can be included in the project. Upon inclusion in the project, a declaration of consent is signed. After this, the patient or with the help of relatives or a health professional will fill in the first questionnaire IPOS-Renal at baseline and then every 6 months. The completed questionnaire is sent by post to primary investigator, or scanned in and sent via e-mail. When 5 months have passed, primary investigator sends a reminder that a new questionnaire must be answered in 1 month (+/- 14 days). This takes place 6, 12, 18 and 24 months after inclusion.

Demographic data will be collected at baseline: age, sex, eGFR, comorbidities, frailty, social conditions, housing conditions, education level, ethnicity and quality of life. Data is collected by principal investigator, who is also responsible for data management. The principal investigator is employed by Department of Renal Medicine at Aarhus University Hospital. Data will be entered and stored in REDCap.

Power calculation Power calculation is based on published data for the hypothesis II, that patients in dialysis treatment have lower mortality than patients on a CKM pathway. Published international data have shown that the hazard ratio (HR) for patients in dialysis treatment compared to patients on a CKM pathway is around 0.5. In a Danish study, the distribution of the patients is seen, thus 90% of patients are in dialysis treatment, while 10% of patients are on a CKM pathway. Internationally, there are studies with patient distributions where up to 60% of the patients are in dialysis treatment, while 40% of the patients are on CKM pathway. This power calculation is based on an assumption of a patient distribution where 80% of patients are in dialysis treatment and 20% of patients are on a CKM pathway. The Danish Nephrology Society finds a mortality of 30% for patients >70 years of age. Based on this, it is calculated that a sample size of a total of 341 patients would provide a power of >80% and could show an HR of 0.5. The project expects to be able to include 341 patients over a period of two years.

Power calculation was also performed for hypothesis I; Patients on a CKM pathway have a greater improvement in their symptom burden measured with IPOS-Renal than patients in dialysis. This hypothesis required a smaller sample size to achieve a power of >80%. The sample size of 341 patients will therefore also be sufficient to be able to identify differences for this hypothesis.

Statistical considerations The statistical analyses will be performed and processed in STATA 17.0. All hypotheses are tested at a significance level of 0.05. Demographic data for baseline characteristics are presented with mean and standard deviation (SD) for continuous data that can be described by a normal distribution. Continuous data, which cannot be described with a normal distribution, are presented with median and interquartile range (IQR). Categorical data is described with number (n) and proportion in percent (%). Scores for primary outcomes are presented with mean and SD if the data is normally distributed. Continuous variables are compared by t-test or Mann-Whitney test. While categorical variables will be compared by chi2 test. Change in symptom burden over time measured by IPOS-Renal will be continuous data collected at 6 months, 12 months, 18 months and 24 months for patients in dialysis treatment and patients on a CKM pathway, respectively. The results of the two different patient groups are then compared by t-test or Mann-Whitney test. A cox proportional hazard regression analysis will be used in relation to calculating the mortality during the follow-up period for the group of patients in dialysis treatment and patients on CKM pathway, respectively.

Critical considerations The study has some methodological limitations. Since data is collected through self-reported questionnaires, there is a risk of information bias, which can be seen in either an over- or under-reporting of symptom burden. We also expect to see a difference between the two patient groups in relation to age, frailty and comorbidity. Attempts will be made to take these differences into account in the statistical analyses. We expect the group of patients in dialysis treatment to be the largest. At the same time, we expect that this group will have a lower mortality and a greater burden of symptoms measured with IPOS-Renal compared to patients on the CKM pathway. On the contrary, we expect that the patients on a CKM pathway have higher mortality and lower symptom burden measured with IPOS-Renal compared to patients on dialysis. The study's strength of 80% is considered a strength for the study, and one must assume that the results found are not based on chance, but contain the real true values.

Ethical considerations Informed written consent will be obtained from all patients prior to the study. Participation in the study will be based on consent to care and treatment in accordance with the health legislation, chapter 5, section 15. According to the Scientific Ethics Committee, it is not required to report the study. This study will be conducted in accordance with the ethical principles of medical research involving human subjects based on the World Medical Association Declaration of Helsinki to protect patients' rights.

On 05.01.2022, the Danish Data Protection Authority has given permission for the registration of sensitive personal data in the research project, Case no. 788266.

Information relating to experimental subjects is protected in accordance with the General Data Protection Regulation and patient rights according to the health legislation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease stage V
* Patients >75 years
* Patients who have decided on future treatment with either dialysis (haemodialysis or peritoneal dialysis) or a CKM pathway

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients eligible for kidney transplantation
* Patients who have decided on home haemodialysis
* Patients who do not wish to participate in the study
* Patients who are unable to participate in the study due to cognitive impairment

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: The patients will be included right after they have made their decision about treatment - dialysis (haemodialysis or peritoneal dialysis) or CKM pathway. In addition, patients must meet inclusion criteria. The patients will be observed for at least two years or until death. The study is expected to start on 15.03.2023, and it is expected to be completed on 15.09.2025.
Sampling Method: Non-Probability Sample
Enrollment: 341 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
IPOS score | after six months, after 12 months, after 18 months and after 24 months
  A score between zero and 40. A high score means a high symptom burden

SECONDARY OUTCOMES:
Mortality | For two years
  Death or a live uptil two years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Finderup, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Renal Medicine, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No